CLINICAL TRIAL: NCT06446765
Title: Mindfulness-based Neurofeedback to Augment Dialectical Behavior Therapy (DBT) for Adults With Borderline Personality Disorder (Aim 1)
Brief Title: Mindfulness-based Neurofeedback to Augment Psychotherapy for Adults With Borderline Personality Disorder
Acronym: MIND-BPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Connecticut Mental Health Center (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000037582; 1R61MH135009-01A1 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Borderline Personality Disorder
Keywords: fMRI neurofeedback; mindfulness
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- mindfulness-based Neurofeedback (Experimental): Participants will participate in one session of mindfulness-based fMRI neurofeedback followed by 20 weeks of remote online weekly Dialectical Behavior Therapy skills group.
  Interventions: Behavioral: mindfulness-based Neurofeedback
- control Neurofeedback (Other): Participants will participate in one session of control fMRI neurofeedback followed by 20 weeks of remote online weekly Dialectical Behavior Therapy skills group.
  Interventions: Other: control Neurofeedback

INTERVENTIONS:
Behavioral: mindfulness-based Neurofeedback — Participants will complete one session of mindfulness-based fMRI neurofeedback prior to 20 weeks of remote online weekly DBT skills group.
  Arms: mindfulness-based Neurofeedback
Other: control Neurofeedback — Participants will complete one session of control fMRI neurofeedback prior to 20 weeks of remote online weekly DBT skills group.
  Arms: control Neurofeedback

SUMMARY:
The purpose of this study is to test the ability of mindfulness-based real time functional magnetic resonance imaging (fMRI) neurofeedback (mbNF) to increase the benefits of evidence-based psychotherapy for adults with Borderline Personality Disorder (BPD).

DETAILED DESCRIPTION:
The focus of this study is Aim 1.

ELIGIBILITY:
Inclusion criteria:

* age 18-60,
* be able to provide written informed consent,
* meet criteria for BPD on semi-structured clinical interview,
* able to plan to keep any prescribed medications and psychotherapy constant during the study
* fluent in English.

Exclusion criteria:

* current DBT psychotherapy outside the study
* lifetime primary psychotic disorder or Bipolar I disorder
* developmental disorder (e.g. autism)
* history of learning disorder
* moderate or severe substance use disorder in the last 6 months
* active suicidal ideation with intent or plan in the past 3 months
* history of major medical or neurologic disorder
* MRI contraindications, including pregnancy
* poor performance on reading task (WRAT > 11 errors)
* newly prescribed medications in the past 8 weeks
* daytime sedating medications (e.g. benzodiazepines, opiates, sedating neuroleptics)
* any scheduled daily benzodiazepines
* change in psychotherapy type or frequency in the past 12 weeks.
* At the discretion of the study PI

Eligibility will be determined by study personnel.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in within-Default Mode Network (DMN) resting state functional connectivity after one session of neurofeedback (NF) | From baseline (immediately before neurofeedback) to immediately after neurofeedback on the same day
  Defined as within-DMN connectivity as the resting state seed-based connectivity between core nodes of medial prefrontal cortex (mPFC) and posterior cingulate cortex (PCC). Change = post-NF within-DMN connectivity - pre-NF within-DMN connectivity.
Change in DMN-Frontoparietal Control Network (FPCN) anticorrelation in resting state functional connectivity data after one session of neurofeedback | From baseline (immediately before neurofeedback) to immediately after neurofeedback on the same day
  Defined as DMN-FPCN anticorrelation as the fMRI seed-based connectivity from mPFC to dorsolateral prefrontal cortex (dlPFC)). Change = post-NF mPFC-dlPFC anticorrelation - pre-NF mPFC-dlPFC anticorrelation

SECONDARY OUTCOMES:
Change from baseline in state mindfulness on State Mindfulness Scale (SMS) score on same day after neurofeedback. | From baseline (immediately before neurofeedback) to immediately after neurofeedback on the same day
  The State Mindfulness Scale (SMS) is a validated self-reported 21 item instrument assessing state mindfulness over the past 15 minutes. Possible scores range from 21 (not mindful) to 105 (very mindful).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Fineberg, MD PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing will occur as required by NIMH through the National Data Archive.

REFERENCES:
- [Derived] Jones KG, Vandewouw MM, Awasthi J, Alario AA, Bauer C, Brewer B, Campbell N, Denning D, Greene KD, Hammoud J, Hinds O, Huffman S, Maerker C, Paprotna S, Qiu M, Swinchoski B, Taylor A, Waite E, Wighton P, Whaley M, Papa J, Gordon KD, Hampson M, Whitfield-Gabrieli S, Fineberg SK. A protocol for MIndfulness-based Neurofeedback to augment DBT psychotherapy for adults with Borderline Personality Disorder (MIND-BPD). medRxiv [Preprint]. 2025 Nov 19:2025.11.18.25340531. doi: 10.1101/2025.11.18.25340531. PMID 41332880